CLINICAL TRIAL: NCT05187455
Title: Pharmacokinetics of Sugammadex for the Reversal of Moderate Neuromuscular Blockade in Patients During Renal Transplantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Collaborators: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, bo xu, associate chief physician, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Renal Transplantation
Record Dates: First submitted 2021-12-03; First posted 2022-01-11 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Pharmacokinetics
Keywords: Sugammadex; renal transplantation
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Renal transplantation(S group) (Experimental): n=17,CLCR≤30ml/min
  Interventions: Drug: Sugammadex
- the control group (Experimental): n=17, CLCR≥80ml/min
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — Each patient received a single dose administration of sugammadex 2mg/kg at reappearance of the second twitch of the train-of-four (TOF).
  Other Names: Org 25969; Bridion

SUMMARY:
The purpose of this study is to illustrate pharmacokinetics of sugammadex in reversal of rocuronium-induced moderate neuromuscular blockade in patients during renal transplantation

DETAILED DESCRIPTION:
34 patients undergoing renal transplantation or elective surgery are divided into 2 groups, including transplantation group (S group,n=17) and control group (C group, n=17). Patients age 18 to 65 and ASA glass I-III

Anaesthesia is induced and maintained with i.v. propofol and an opioid. Neuromuscular monitoring was performed at the adductor pollicis muscle with acceleromyography (TOF-Watch®SX, Organon Ireland Ltd, a division of Merck and Co., Dublin, Ireland). After calibration of the TOF-Watch®SX, an i.v. bolus dose of rocuronium 0.6 mg/kg is given for tracheal intubation, with maintenance doses 0.15mg/kg if T2 reappears to maintain moderate NMB Patients receive sugammadex 2 mg/kg i.v. for reversal when surgery finish and T2 reappears.

Venous blood samples of C group(within 12hours) and S group(within 48hours) are obtained before administration of Sug and at specified time points after administration of Sug to determine plasma concentration using HPLC-MS. Time from start of administration of Sug to recovery of TOF ratio to 0.7, 0.8, 0.9 and other clinical indicators are also recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergo emergency renal transplantation under general anesthesia(CLCR≤30ml/min),or patients undergo elective surgery in supine position(CLCR≥80ml/min)
2. Patients age 18 to 65
3. ASA glass I-III

Exclusion Criteria:

1. patients suffering obstructive sleep apnea hypopnea syndrome or BMI≥28kg/m2
2. Pregnant or lactating women
3. neuromuscular disorders, hepatic dysfunction, cardiac disease, a history of malignant hyperthermia, or
4. allergic history during general anesthesia
5. patients receiving aminoglycoside antibiotics, anticonvulsants, magnesium,fusidic acid,toremifene and/or flucloxacillin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Plasma Concentration of Sugammadex | Samples were obtained pre-dose and at specified post-dose time points. C group: up to 12 hours post-dose, S group: up to 48 hours post-dose
  venous blood samples were obtained

SECONDARY OUTCOMES:
Recovery Time and TOF ratio | up to 10 minutes from start of sugammadex
  Time from start of administration of sugammadex to recovery of the T4/T1 Ratio to 0.7 、0.8、0.9
Adverse Event | Up to 2 days
  Percentage of Participants With ≥1 Adverse Event

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Hospital of Traditional Chinese Medicine, Guanzhou, Guangdong, China

REFERENCES:
- [Background] McDonagh DL, Benedict PE, Kovac AL, Drover DR, Brister NW, Morte JB, Monk TG. Efficacy, safety, and pharmacokinetics of sugammadex for the reversal of rocuronium-induced neuromuscular blockade in elderly patients. Anesthesiology. 2011 Feb;114(2):318-29. doi: 10.1097/ALN.0b013e3182065c36. PMID 21239968
- [Background] Panhuizen IF, Gold SJ, Buerkle C, Snoeck MM, Harper NJ, Kaspers MJ, van den Heuvel MW, Hollmann MW. Efficacy, safety and pharmacokinetics of sugammadex 4 mg kg-1 for reversal of deep neuromuscular blockade in patients with severe renal impairment. Br J Anaesth. 2015 May;114(5):777-84. doi: 10.1093/bja/aet586. Epub 2015 Mar 31. PMID 25829395
- [Background] Adams DR, Tollinche LE, Yeoh CB, Artman J, Mehta M, Phillips D, Fischer GW, Quinlan JJ, Sakai T. Short-term safety and effectiveness of sugammadex for surgical patients with end-stage renal disease: a two-centre retrospective study. Anaesthesia. 2020 Mar;75(3):348-352. doi: 10.1111/anae.14914. Epub 2019 Nov 12. PMID 31721151
- [Background] de Souza CM, Tardelli MA, Tedesco H, Garcia NN, Caparros MP, Alvarez-Gomez JA, de Oliveira Junior IS. Efficacy and safety of sugammadex in the reversal of deep neuromuscular blockade induced by rocuronium in patients with end-stage renal disease: A comparative prospective clinical trial. Eur J Anaesthesiol. 2015 Oct;32(10):681-6. doi: 10.1097/EJA.0000000000000312. PMID 26225497